CLINICAL TRIAL: NCT04398420
Title: Safety and Efficacy of TVERP in BPH Patients With Prostate Size ˃30 and ≤80 ml: a Comparison Study Between TVERP With the Plasma Vaporisation Button, Bipolar TURis and HoLEP Treatments.
Brief Title: Transurethral Vapor Enucleation Resection of the Prostate (TVERP), Bipolar TURis and HoLEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low recruitment. FUP of enrolled patients will be performed until LPLV.
Sponsor: Olympus Surgical Technologies Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVERP01
Record Dates: First submitted 2020-05-12; First posted 2020-05-21 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Benign Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TVERP (Active Comparator)
  Interventions: Device: TVERP
- TURis (Active Comparator)
  Interventions: Device: TURis
- HoLEP (Active Comparator)
  Interventions: Device: HoLEP

INTERVENTIONS:
Device: TVERP — Transurethral Vapor Enucleation Resection of the prostate
  Arms: TVERP
Device: TURis — Transurethral Vapor Enucleation Resection of the prostate
  Arms: TURis
Device: HoLEP — Transurethral Vapor Enucleation Resection of the prostate
  Arms: HoLEP

SUMMARY:
To verify the safety and efficacy of the use of the plasma vaporisation button in Transurethral Vapor Enucleation and Resection of the prostate (TVERP) for treatment of Benign prostatic hypertrophy (BPH) patients with prostate ˃30 and ≤80 ml compare to TURis or HoLEP surgery methods.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age older than 22 and younger than 75 years of age
2. The patient should be a candidate for surgical treatment of bladder outlet obstruction.
3. Patients with BPH and surgical indication (refractory to medical treatment, refractory or recurrent urinary retention, recurrent haematuria, bladder stones, recurrent infections, hydronephrosis)
4. Prostate volume ˃30 and ≤80 ml
5. PSA <4 ng/ml in patients above 55 years old and a prostate cancer risk less than 35%. (Prostate cancer risk calculator).
6. IPSS ≥8 (moderate to severe)
7. Indications for TURIS
8. maximum urinary flow (Qmax) <10ml/second
9. A written informed consent signed by the patient (including patient's agreement to randomization and treatment).

Exclusion Criteria:

1. Patients under anti-inflammatory or steroid therapy
2. Patients under anti-coagulation at a level that could be exposed to a very high risk of complications based on a comprehensive pre-operatory evaluation.
3. Renal insufficiency Serum creatinine (Scr) >1.5 x upper limit of normal (ULN); AST and ALT>2.5 x ULN;Total bilirubin >1.5 x ULN
4. Previous neurogenic lower urinary tract dysfunction.
5. Patients with urethral strictures
6. Severe pulmonary disease and cardio-vascular disorder 、Coagulopathy，and contraindications to anesthesia and surgery.
7. Concurrent participation in any other clinical study
8. Any of the following within the 12 months prior to study: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
9. Previous bladder outlet surgery.
10. A clinically significant acute illness.
11. Intake of medication in which the principle investigator considers to preclude enrollment into the trial.
12. Known disease of the central or peripheral nervous system.
13. Any clinical evidence of carcinoma of the prostate.
14. HIV positive or any other immunosuppressive disorder.
15. Psychological/psychiatric disease /Known cognitive disorder.

Ages: 22 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
change of blood level | Measurement of pre-operative and immediate post-operative period (6 hours and 24 hours) hemoglobin and hematocrit levels will be performed.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Renmin Hospital,Wuhan University, Wuhan, Hubei
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang